CLINICAL TRIAL: NCT00696774
Title: Attributes of Response in Depressed Patients Switched to Treatment With Duloxetine (ARDENT Study)
Brief Title: Switching to Duloxetine in Patients With Depression
Acronym: ARDENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12349; F1J-CR-S022 (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2010-08-11 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (Experimental): Patients who met criteria in Study Period I (screening) were treated with duloxetine 60 milligrams (mg) once daily (QD) in an open-label manner for 4 weeks (Study Period II). Study Period II was considered the acute therapy period. Study Period III was a 4-week interval where patients who did not respond during Study Period II had their duloxetine doses optimized to 120 mg.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Study Period II (Acute Therapy): 60 mg capsules, QD, for 4 weeks.
  Study Period III (Optimization): Responder group - 60 mg capsules, QD, for 4 weeks more. Non-responder group - 120 mg capsules, QD, for 4 weeks more.
  Other Names: LY248686; Cymbalta

SUMMARY:
The purpose of this study is to help answer the following research question: Whether switching to duloxetine improves depressed mood when current treatment did not work well for patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 18 years or older who meet criteria for Major Depressive Disorder (MDD).
* Currently receiving a selective serotonin reuptake inhibitor (SSRI) or a serotonin-norepinephrine reuptake inhibitor (SNRI) class of antidepressant for at least a month for the treatment of depression.
* Females of child-bearing potential (not surgically sterilized and between menarche and 1 year postmenopause) to test negative for pregnancy based on a urine pregnancy test and to agree to use a reliable method of birth control.

Exclusion Criteria:

* Women who are pregnant or plan to be pregnant or are breastfeeding.
* To have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication.
* Diagnosed with treatment resistant depression.
* History of bipolar disorder, schizophrenia, or other psychotic disorders.
* To have previously taken duloxetine that didn't work.
* Judged to be at serious suicidal risk in the opinion of the investigator and/or score >=3 on Item 3 (suicide) of the 17-Item Hamilton Depression Rating Scale (HAMD-17) at screening (Visit 1) or baseline (Visit 2).
* A serious medical illness that may need treatment during the study.
* Taking certain medications that are not allowed in this study.
* To have a history of alcohol and/or drug abuse or dependence within the past year.
* To have uncontrolled narrow-angle glaucoma.
* To have allergic reactions to many medicines.
* To have undergone "shock" therapy (Electroconvulsive Therapy) or "magnet" treatment (Transcranial Magnetic Stimulation) within the past year.
* To initiate "talk therapy" (psychotherapy) just before or during the study.
* To have chronic pain and you have been taking medicine for it for the last 6 months.
* To have certain liver diseases.
* To have kidney disease or undergoing dialysis.
* Abnormal thyroid stimulating hormone (TSH) concentration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guri-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 270 participants began the study. 26 were screen failures (17 did not meet entry criteria, 7 decided to withdraw, and 2 withdrew based on the physician's decision). 2 participants discontinued before enrollment (1 was lost to follow-up and 1 decided to withdraw).
Groups:
- Responders: 60 milligram (mg) duloxetine capsules, once daily (QD), for 4 weeks (Study Period II). Responder group - 60 mg capsules, QD, for 4 weeks more (Study Period III).
- Non-Responders: 60 mg duloxetine capsules, QD, for 4 weeks (Study Period II). Non-Responder group - 120 mg capsules, QD, for 4 weeks more (Study Period III).
- Unclassified: Participants who received 60 milligram (mg) duloxetine capsules, once daily (QD), for 4 weeks (Study Period II) with unknown response status.
Period: Period II
Arm/Group | Responders | Non-Responders | Unclassified
Started | 115 | 91 | 36 (1 participant did not receive study drug and was not included in the safety analyses.)
Completed | 115 | 91 | 0
Not Completed | 0 | 0 | 36
Not completed — Adverse Event | 0 | 0 | 15
Not completed — Lost to Follow-up | 0 | 0 | 4
Not completed — Protocol Violation | 0 | 0 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Sponsor Decision | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2
Period: Period III
Arm/Group | Responders | Non-Responders | Unclassified
Started | 113 (115 reported at Week 4; 113 started Period 3 (1 lost to follow-up and 1 protocol violation).) | 88 (91 reported at Week 4; 88 start Period 3 (1 adverse event, 1 protocol violation, 1 lack of efficacy)) | 0
Completed | 106 | 81 (82 participants were reported at Week 8; 81 completed Week 8 as 1 participant decided to withdraw.) | 0
Not Completed | 7 | 7 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Sponsor Decision | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Duloxetine Responders: 60 milligram (mg) duloxetine capsules, once daily (QD), for 4 weeks (Study Period II). Responder group - 60 mg capsules, QD, for 4 weeks more (Study Period III).
- Duloxetine Non-Responders: 60 mg duloxetine capsules, QD, for 4 weeks (Study Period II). Non-responder group - 120 mg capsules, QD, for 4 weeks more (Study Period III).
- Total: Total of all reporting groups
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders | Unclassified | Total
Number analyzed (Participants) | 115 | 91 | 36 | 242
Age Continuous [Mean (Standard Deviation); unit: years] | 43.5 (12.9) | 45.6 (12.5) | 47.4 (10.6) | 44.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 64 | 30 | 182
  Male | 27 | 27 | 6 | 60
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 67 | 66 | 17 | 150
  East Asian | 43 | 23 | 12 | 78
  African | 1 | 0 | 2 | 3
  Hispanic | 2 | 2 | 3 | 7
  West Asian | 2 | 0 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 18 | 11 | 9 | 38
  Brazil | 9 | 11 | 13 | 33
  China | 25 | 13 | 3 | 41
  Canada | 63 | 56 | 11 | 130
Had Major Depressive Disorder (MDD) Hospitalizations in the Past 24 Months [Number; unit: participants]
  Yes | 8 | 5 | 2 | 15
  No | 107 | 86 | 34 | 227
Had Previous MDD in the Past 24 Months [Number; unit: participants]
  Yes | 79 | 54 | 24 | 157
  No | 36 | 37 | 12 | 85
Had at Least One Historical Illness [Number; unit: participants]
  Yes | 44 | 32 | 15 | 91
  No | 71 | 59 | 21 | 151
Previous Treatment [Number; unit: participants] — Previous selective serotonin reuptake inhibitor (SSRI) or serotonin norepinephrine reuptake inhibitor (SNRI) treatment.
  participants
    SSRI | 83 | 69 | 25 | 177
    SNRI | 31 | 21 | 9 | 61
    Missing or Unknown | 1 | 1 | 2 | 4
17-Item Hamilton Depression Rating Scale (HAMD-17) Anxiety/Somatization Score [Mean (Standard Deviation); unit: units on a scale] — The Anxiety/Somatization Subscale (Items 10-13, 15, 17) evaluates severity of psychic and somatic manifestations of anxiety as well as agitation. Total subscale scores range from 0 (normal) to 18 (severe).
  units on a scale | 7.7 (2.1) | 8.0 (2.0) | 7.4 (1.7) | 7.8 (2.0)
17-Item Hamilton Depression Rating Scale (HAMD-17) Core Score [Mean (Standard Deviation); unit: units on a scale] — The Core subscale (Items 1,2,3,7,8) evaluates "core" symptoms of depression. Total subscale scores range from 0 (normal) to 20 (severe).
  units on a scale | 8.1 (2.6) | 9.0 (2.6) | 7.9 (2.8) | 8.4 (2.7)
17-Item Hamilton Depression Rating Scale (HAMD-17) Maier Score [Mean (Standard Deviation); unit: units on a scale] — The Maier subscale (Items 1,2,7,8,9,10) represents the "core" symptoms of depression. Total subscale scores range from 0 (normal) to 24 (severe).
  units on a scale | 10.7 (2.6) | 11.7 (2.6) | 10.0 (2.7) | 11.0 (2.7)
17-Item Hamilton Depression Rating Scale (HAMD-17) Retardation Score [Mean (Standard Deviation); unit: units on a scale] — The Retardation Subscale (Items 1,7,8,14) evaluates dysfunction in mood, work, and sexual activity, as well as overall motor retardation. Total subscale scores range from 0 (normal) to 14 (severe).
  units on a scale | 7.1 (2.1) | 8.2 (1.9) | 7.2 (2.4) | 7.5 (2.1)
17-Item Hamilton Depression Rating Scale (HAMD-17) Sleep Score [Mean (Standard Deviation); unit: units on a scale] — The Sleep Subscale (Items 4,5,6) evaluates initial, middle, and late insomnia. Total subscale scores range from 0 (no difficulty) to 6 (difficulty).
  units on a scale | 3.1 (1.6) | 3.4 (1.4) | 3.2 (1.7) | 3.2 (1.5)
17-Item Hamilton Depression Rating Scale (HAMD-17) Total Score [Mean (Standard Deviation); unit: units on a scale] — The HAMD-17 measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
  units on a scale | 21.3 (4.5) | 23.3 (4.5) | 20.7 (4.5) | 21.9 (4.6)
Age of First Episode of MDD [Mean (Standard Deviation); unit: years] | 35.2 (11.7) | 33.5 (13.6) | 36.9 (12.8) | 34.8 (12.6)
Brief Pain Inventory - Short Form (BPI-SF) Average Pain Score [Mean (Standard Deviation); unit: Units on a scale] — A self-reported scale that measures the severity of pain based on the average pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  Units on a scale | 4.7 (1.9) | 5.0 (2.0) | 4.4 (2.2) | 4.8 (2.0)
Brief Pain Inventory - Short Form Interference Score [Mean (Standard Deviation); unit: Units on a scale] — The BPI-SF interference score asks about the degree to which pain interferes with mood, walking and other physical activity, work, social activity, relations with others, and sleep. BPI-SF interference score ranges from 0 (no interference) to 10 (interferes completely).
  Units on a scale | 5.2 (1.6) | 5.9 (1.8) | 5.2 (1.9) | 5.5 (1.8)
Changes in Sexual Function Questionnaire (CSFQ) [Mean (Standard Deviation); unit: Units on a scale] — A 14-item patient-rated scale designed to assess medication-related changes in sexual activity/functioning. Items are rated from 1 (never, low enjoyment or pleasure) to 5 (every day/great enjoyment or pleasure). CSFQ measures 5 dimensions of sexual behavior: pleasure; desire/frequency; desire/interest; arousal; orgasm. CSFQ total score is obtained across all 5 dimensions. Lower scores are associated with sexual dysfunction/diminished sexual functioning. Total scores <=47 (men) and <=41 (women) indicate global sexual dysfunction, with all phases of the sexual response cycle being affected.
  Units on a scale | 35.3 (10.3) | 35.4 (9.8) | 33.8 (9.4) | 35.1 (10.0)
Clinical Global Impressions - Severity (CGI-Severity) Score [Mean (Standard Deviation); unit: Units on a scale] — Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  Units on a scale | 4.2 (0.6) | 4.4 (0.6) | 4.3 (0.7) | 4.3 (0.6)
Duration of the Current Episode [Mean (Standard Deviation); unit: days] | 249.4 (378.3) | 264.5 (318.1) | 194.1 (182.6) | 247.3 (333.3)
Hamilton Anxiety Rating Scale (HAMA) Total Score [Mean (Standard Deviation); unit: Units on a scale] — The HAMA scale measures anxiety symptoms accompanying major depressive disorder (MDD). Each item of the 14-item HAMA was scored from 0 (not present) to 4 (very severe), with a resulting maximum total score of 56.
  Units on a scale | 17.9 (6.8) | 21.4 (6.8) | 17.9 (7.6) | 19.2 (7.1)
Number of MDD Hospitalizations in the Past 24 Months [Mean (Standard Deviation); unit: hospitalizations] | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0)
Number of Previous MDD Episodes in the Past 24 Months [Mean (Standard Deviation); unit: MDD episodes] | 1.6 (0.8) | 1.5 (0.7) | 1.8 (1.5) | 1.6 (0.9)
Sheehan Disability Scale (SDS) [Mean (Standard Deviation); unit: Units on a scale] — The SDS is completed by the patient and is used to assess the effect of the patient's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the patient's work/social/family life.
  Units on a scale | 5.4 (2.9) | 6.3 (3.0) | 5.5 (3.0) | 5.7 (3.0)
Treatment Satisfaction Questionnaire for Medication (TSQM) [Mean (Standard Deviation); unit: Units on a scale] — The TSQM is a participant-reported measure that best describes how the study medication makes them feel since the last study visit, assessing perceived effectiveness, severity of side effects, and convenience. Convenience, Effectiveness, Side-Effects, and Global Satisfaction scale scores range from 0 (extremely dissatisfied) to 100 (extremely satisfied).
  Units on a scale | 44.2 (17.6) | 41.6 (18.2) | 47.2 (20.8) | 43.7 (18.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Brief Pain Inventory-Modified Short Form (BPI-SF) Interference Score Between Responder and Non-Responder Participants at 4 Weeks
Description: BPI-SF interference score asks about the degree to which pain interferes with mood, walking and other physical activity, work, social activity, relations with others, and sleep. BPI-SF interference score ranges from 0 (no interference) to 10 (interferes completely). Response is defined as a >=50% reduction in the Maier subscale score from baseline. The Maier subscale (Items 1,2,7,8,9,10) represents "core" symptoms of depression. Total subscale scores range from 0 (normal) to 24 (severe). Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 4 weeks
Population: Efficacy Population: Participants who had at least one post-baseline observation were included in the efficacy analysis. The group "Unclassified" was excluded from statistical testing.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale | -2.35 [-2.83 to -1.87] | -1.69 [-2.18 to 1.21]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Test type: Superiority or Other; p = 0.005, Adjusted Repeated Measures Analysis; Model terms: baseline score & CGI, age, sex, country, prev treatment, prev treatment discontinuation reason, response group, visit & response-by-visit; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.12 to -0.20] — Least Squares Mean Difference = Responders - Non-Responders

2. Secondary Outcome: Percentage of Participants Meeting Criteria for Response on the 17-Item Hamilton Depression Rating Scale (HAMD-17) Maier Subscale at 4 and 8 Weeks
Description: The Maier subscale (Items 1,2,7,8,9,10) represents the "core" symptoms of depression. Total subscale scores range from 0 (normal) to 24 (severe). Response is defined as a >=50% reduction in the Maier subscale score from baseline.
Time Frame: Baseline, 4 weeks, 8 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Duloxetine: 60 milligram (mg) duloxetine capsules, once daily (QD), for 4 weeks. Responder group - 60 mg capsules, QD, for 4 weeks more. Non-responder group - 120 mg capsules, QD, for 4 weeks more.
Arm/Group | Duloxetine
Number analyzed (Participants) | 193
Percentage of participants
  Week 4 (n=193) | 56.0 [48.7 to 63.1]
  Week 8 (n=179) | 73.7 [66.7 to 80.0]

3. Secondary Outcome: Change From Baseline HAMD-17 Total Score at 8 Weeks
Description: The HAMD-17 total score measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe). Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale | -15.64 [-16.86 to -14.41] | -9.79 [-11.10 to -8.47]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.85, 95% CI 2-sided [-7.34 to -4.36] — Least Squares Mean Difference = Responders - Non-Responders

4. Secondary Outcome: Change From Baseline HAMD-17 Core Subscale at 8 Weeks
Description: The Core subscale (Items 1,2,3,7,8) evaluates "core" symptoms of depression. Total subscale scores range from 0 (normal) to 20 (severe). Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale | -6.87 [-7.41 to -6.33] | -4.40 [-4.99 to -3.81]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.47, 95% CI 2-sided [-3.13 to -1.81] — Least Squares Mean Difference = Responders - Non-Responders

5. Secondary Outcome: Change From Baseline HAMD-17 Maier Subscale at 8 Weeks
Description: The Maier subscale (Items 1,2,7,8,9,10) represents the "core" symptoms of depression. Total subscale scores range from 0 (normal) to 24 (severe). Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale | -8.58 [-9.25 to -7.90] | -5.29 [-6.01 to -4.56]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.29, 95% CI 2-sided [-4.10 to -2.48] — Least Squares Mean Difference = Responders - Non-Responders

6. Secondary Outcome: Change From Baseline HAMD-17 Anxiety/Somatization Subscale at 8 Weeks
Description: The Anxiety/Somatization Subscale (Items 10-13, 15, 17) evaluates severity of psychic and somatic manifistations of anxiety as well as agitation. Total subscale scores range from 0 (normal) to 18 (severe). Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale | -5.29 [-5.84 to -4.73] | -3.07 [-3.68 to -2.47]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.22, 95% CI 2-sided [-2.89 to -1.54] — Least Squares Mean Difference = Responders - Non-Responders

7. Secondary Outcome: Change From Baseline HAMD-17 Retardation/Somatization Subscale at 8 Weeks
Description: The Retardation Subscale (Items 1,7,8,14) evaluates dysfunction in mood, work, and sexual activity, as well as overall motor retardation. Total subscale scores range from 0 (normal) to 14 (severe). Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale | -5.51 [-5.98 to -5.05] | -3.63 [-4.14 to -3.13]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-2.45 to -1.30] — Least Squares Mean Difference = Responders - Non-Responders

8. Secondary Outcome: Change From Baseline HAMD-17 Sleep Subscale at 8 Weeks
Description: The Sleep Subscale (Items 4,5,6) evaluates initial, middle, and late insomnia. Total subscale scores range from 0 (no difficulty) to 6 (difficulty). Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale | -2.27 [-2.59 to -1.96] | -1.31 [-1.64 to -0.97]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-1.31 to -0.63] — Least Squares Mean Difference = Responders - Non-Responders

9. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Rating Scale (HAMA) at 8 Weeks
Description: The HAMA scale measures anxiety symptoms accompanying major depressive disorder (MDD). Each item of the 14-item HAMA was scored from 0 (not present) to 4 (very severe), with a resulting maximum total score of 56. Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale | -12.97 [-14.37 to -11.56] | -8.55 [-10.04 to -7.06]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.42, 95% CI 2-sided [-6.04 to -2.80] — Least Squares Mean Difference = Responders - Non-Responders

10. Secondary Outcome: Change From Baseline in the Clinical Global Impression - Severity (CGI-Severity) Scale at 8 Weeks
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale | -2.52 [-2.75 to -2.30] | -1.40 [-1.65 to -1.14]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-1.42 to -0.84] — Least Squares Mean Difference = Responders - Non-Responders

11. Secondary Outcome: Change From Baseline in the Brief Pain Inventory - Modified Short Form (BPI-SF) Average Pain Score at 8 Weeks
Description: A self-reported scale that measures the severity of pain based on the average pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale | -2.56 [-3.13 to -1.99] | -2.14 [-2.75 to -1.53]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.08 to -0.24] — Least Squares Mean Difference = Responders - Non-Responders

12. Secondary Outcome: Change From Baseline in Patient Global Impression - Improvement (PGI-I) Scale Score at 8 Weeks
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse). Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale | 2.12 [1.85 to 2.38] | 2.61 [2.33 to 2.90]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.81 to -0.18] — Least Squares Mean Difference = Responders - Non-Responders

13. Secondary Outcome: Change From Baseline in the Sexual Functioning Questionnaire Clinical Version (CSFQ) at 4 and 8 Weeks
Description: A 14-item patient-rated scale assesses medication-related changes in sexual activity/functioning. Items rated from 1 (never, low enjoyment/pleasure) to 5 (every day, great enjoyment/pleasure). CSFQ measures 5 dimensions of sexual behavior: pleasure; desire/frequency; desire/interest; arousal; orgasm. Lower total scores are associated with diminished sexual functioning. Total scores <=47 (men) and <=41 (women) indicate global sexual dysfunction, with all phases of sexual response cycle affected. Factors used for adjustment for least squares means are in 'Other relevant information' section.
Time Frame: Baseline, 4 Weeks, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale
  Week 4 | 0.03 [-1.84 to 1.90] | -0.78 [-2.76 to 1.21]
  Week 8 | 1.08 [-0.90 to 3.05] | -0.29 [-2.42 to 1.84]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Week 4; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [-0.99 to 2.60] — Least Squares Mean Difference = Responders - Non-Responders
Statistical Analysis 2: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Week 8; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.36, 95% CI 2-sided [-0.69 to 3.42] — Least Squares Mean Difference = Responders - Non-Responders

14. Secondary Outcome: Change From Baseline in the Treatment Satisfaction Questionnaire for Medication (TSQM) at 4 and 8 Weeks
Description: The TSQM is a participant-reported measure that best describes how the study medication makes them feel since the last study visit, assessing perceived effectiveness, severity of side effects, and convenience. Convenience, Effectiveness, Side-Effects, and Global Satisfaction scale scores range from 0 (extremely dissatisfied) to 100 (extremely satisfied). Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 4 weeks, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale
  Week 4 | 17.64 [12.88 to 22.39] | 2.59 [-2.16 to 7.34]
  Week 8 | 18.67 [13.37 to 23.97] | 8.19 [2.65 to 13.73]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Week 4; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 15.05, 95% CI 2-sided [10.63 to 19.47] — Least Squares Mean Difference = Responders - Non-Responders
Statistical Analysis 2: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Week 8; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 10.48, 95% CI 2-sided [4.72 to 16.24] — Least Squares Mean Difference = Responders - Non-Responders

15. Secondary Outcome: Change From Baseline in the Sheehan Disability Scale (SDS) at 4 and 8 Weeks
Description: The SDS is completed by the patient and is used to assess the effect of the patient's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the patient's work/social/family life. Factors used for adjustment for least squares means are listed in 'Other relevant information' section.
Time Frame: Baseline, 4 weeks, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders
Number analyzed (Participants) | 108 | 85
Units on a scale
  Week 4 | -8.38 [-10.26 to -6.50] | -2.49 [-4.42 to -0.57]
  Week 8 | -9.95 [-11.91 to -7.99] | -5.36 [-7.40 to -3.32]
Statistical Analysis 1: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Week 4; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.88, 95% CI 2-sided [-7.75 to -4.02] — Least Squares Mean Difference = Responders - Non-Responders
Statistical Analysis 2: Comparison: Duloxetine Responders vs Duloxetine Non-Responders; Week 8; Test type: Superiority or Other; Adjusted Repeated Measures Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.59, 95% CI 2-sided [-6.65 to -2.54] — Least Squares Mean Difference = Responders - Non-Responders

ADVERSE EVENTS:
Groups:
- Duloxetine Responders: 60 mg duloxetine capsules, QD, for 4 weeks (Study Period II). Responder group - 60 mg capsules, QD, for 4 weeks more (Study Period III).
Arm/Group | Duloxetine Responders | Duloxetine Non-Responders | Unclassified
Serious Adverse Events (participants affected / at risk) | 0/115 | 2/91 | 0/35
Other Adverse Events (participants affected / at risk) | 71/115 | 59/91 | 22/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine Responders (N=115) | Duloxetine Non-Responders (N=91) | Unclassified (N=35)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine Responders (N=115) | Duloxetine Non-Responders (N=91) | Unclassified (N=35)
Vision blurred (Eye disorders) | 0 (0) | 5 (5) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 13 (13) | 9 (9) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 12 (12) | 14 (14) | 0 (0)
Nausea (Gastrointestinal disorders) | 20 (20) | 15 (15) | 7 (7)
Asthenia (General disorders) | 1 (1) | 2 (2) | 2 (2)
Fatigue (General disorders) | 3 (3) | 7 (7) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (5) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 15 (15) | 10 (10) | 5 (5)
Headache (Nervous system disorders) | 15 (15) | 15 (15) | 2 (2)
Somnolence (Nervous system disorders) | 8 (8) | 7 (7) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 6 (6) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (10) | 10 (10) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 2 (2)
Hot flush (Vascular disorders) | 3 (3) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days